CLINICAL TRIAL: NCT05232734
Title: CaffeinICU Study - A Multi-centre Pilot Study to Examine the Safety and Feasibility of Oral Caffeine in Critically Ill Adult Patients With Low Glasgow Coma Scale Score.
Brief Title: CaffeinICU Study - A Study on Oral Caffeine in ICU Patients With Coma
Acronym: CaffeinICU
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study amendment done in view of low recruitment numbers. Updated HSA approved study protocol awaiting IRB approval before study re-commences
Sponsor: Singapore General Hospital (Other)
Collaborators: Sengkang General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/2556
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Depressed GCS
Keywords: Caffeine; Depressed GCS; Mechanical Ventilation
MeSH Terms: interventions — caffeine citrate; Solutions; Caffeine

STUDY DESIGN:
Intervention Model Description: Multi-center pilot observational single-arm clinical feasibility trial
Masking Description: The study drug is oral caffeine solution which will be prepared by pharmacy laboratory using caffeine powder into 20mg/mL caffeine solution. The solution will be packed in amber glass bottle ready for administration by nurses at bedside without further dilution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral caffeine group (Experimental): Patients in this arm will receive treatment with oral caffeine
  Interventions: Drug: Caffeine Citrate 20 MG/ML Oral Solution

INTERVENTIONS:
Drug: Caffeine Citrate 20 MG/ML Oral Solution — Caffeine syrup will be prepared by pharmacy laboratory and kept refrigerated (2-8C), to be used within 1 month from the date of preparation by pharmacy laboratory.
  Other Names: Caffeine

SUMMARY:
Background:

Depressed Glasgow Coma Scale (GCS) is common among critically ill patient s in the intensive care unit (ICU). It is one of the main reasons that hampers liberation from mechanical ventilation among ICU patients. Caffeine is commonly used in neonates for the treatment of apnea of prematurity. However, its efficacy has not been established in adult population.

Objective:

To find out the efficacy of oral caffeine in shortening duration of mechanical ventilation among adult patients.

Hypothesis:

Oral caffeine is effective as a central nervous system stimulant among adult patients with depressed GCS.

Study design:

Multi-center, randomised, double blind, placebo controlled clinical trial

Population:

Adult patients (≥ 21 years old) with GCS ≤ 8 from any causes (excluding surgically reversible causes) requiring continuation of mechanical ventilation, whom acute medical issues are stable or has resolved but not suitable for extubation solely due to depressed GCS, not planned for any surgical procedures within 24 hours and not on sedative agents for at least 24 hours, will be included in this study. For patients with primary Central Nervous System (CN lesions, neurologist or neurosurgeon approval will be obtained prior to recruitment. The exclusion criteria include known allergy or adverse reactions from caffeine, pregnant women, breast-feeding women, uncontrolled cardiac arrhythmias, uncontrolled hypertension, hyperactive delirium, patients with chronic kidney disease (CKD, any stage) who received midazolam or morphine infusion, patients who received barbiturate coma, patients who are on theophylline, aminophylline or psychotropic agents at the point of screening for recruitment, patients with feed intolerant, short bowel syndrome and active seizures.

Intervention:

Oral caffeine citrate 5mg/kg/dose twice a day (8am, 2pm) vs placebo

Outcomes:

Primary - Duration of mechanical ventilation Secondary - ICU mortality, 30-days mortality, ICU length of stay, blood pressure, heart rate, incidence of arrhythmia, GCS, incidence of re-intubation and need for tracheostomy

DETAILED DESCRIPTION:
Depressed Glasgow Coma Scale (GCS) is common among critically ill patients in the intensive care unit (ICU). It is one of the main reasons that hampers liberation from mechanical ventilation among ICU patients. Current management of this disorder focuses mainly on supportive care and treatment of the underlying disease. Directed therapies targeting neurochemical and neurotransmitter pathways are not currently available and it represents an important area of research. Caffeine is commonly used in neonates for the treatment of apnea of prematurity. It is a CNS stimulant that stimulates central respiratory drive, increases medullary respiratory center sensitivity to carbon dioxide and improves diaphragmatic contractility. However, its efficacy has not been established in adult population.

Hypothesis:

1. Oral caffeine is safe for use for adult ICU patients with depressed GCS at the selected dose.
2. It is feasible to recruit the stipulated study population from SGH and SKH within the time frame of the study.

Objective:

The primary objectives of the study are:

1. To study the safety of oral caffeine among critically ill adult patients. Specifically, the investigators will observe for changes in the blood pressure and heart rate, as well as any incidence of arrthythmia among critically ill adult patients administered with oral caffeine
2. To study the feasibility of the study. Specifically, the investigators will observe and examine factors and challenges (such as from the inclusion/exclusion criteria, caregiver's willingness to participate) that influence recruitment
3. To estimate the duration of mechanical ventilation with the use of oral caffeine (dose: 5mg/kg/dose twice daily) in adult patients who are critically ill.

The secondary objectives are:

(To describe the ICU mortality, 30-days mortality, ICU length of stay, GCS, incidence of re-intubation, incidence of terminal extubation and need for tracheostomy among critically ill adult patients administered with oral caffeine

Proposed Trial Design:

The investigators propose a pilot multi-center, single arm trial of 10 patients with depressed GCS, assigned to receive oral caffeine. 10 subjects from SGH and SKH who are on mechanical ventilation with depressed GCS will be recruited into this study. No randomisation or blinding will be carried out in this study.

Planned Trial Interventions:

Participants will receive oral caffeine through their feeding tube, 5mg/kg/dose twice daily. Oral caffeine solution (colorless and odorless) will be prepared by pharmacy laboratory and supplied in amber glass bottle. Potential drug-drug interaction with oral caffeine will be monitored throughout the study period:

1. CYP1A2 enzyme inhibitors and inducers to be taken with caution/prohibited
2. CYP1A2 substrates to be taken with caution/prohibited

Screening Visits and Procedures:

Study subjects will be identified through referral by the attending ICU medical team or weekly patient screening. Potential subjects will be reviewed by one of the study team members for recruitment eligibility, according to the study inclusion and exclusion criteria. Consent will be obtained from patient's Legally Appointed Representative(LAR) if available, or the next of kin within 72 hours.

Duration of follow up:

Patient clinical status will be monitored on daily basis until 30 days after recruitment or discharge from hospital, whichever earlier.

Data collection:

Data collection will be done prospectively. All parameters collected are part of standard of care, no additional test required for the purpose of this study. Study feasibility data will be collected from screening and recruitment logs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 21 years old),
2. Patients with encephalopathy (GCS ≤ 8) limiting extubation, where encephalopathy is deemed by clinician to be unresponsive to treatment or not eligible for treatment to reverse the encephalopathy (eg. transplantation) or if no treatment exists, and
3. Patients who are not planned for any surgical procedures within 24 hours
4. Patients who are not on sedative agents for at least 24 hours (exception for low dose fentanyl of up to 30mcg/h and dexmedetomidine of up to 0.5mcg/kg/h for analgesia/sedation/tube tolerance)

   * For patients with primary CNS lesions, neurologist or neurosurgeon approval will be obtained prior to recruitment.

Exclusion Criteria:

1. Known allergy or adverse reactions from caffeine,
2. Pregnant women,
3. Breast-feeding women,
4. Patients with uncontrolled cardiac arrhythmias,
5. Patients with uncontrolled hypertension,
6. Patients with hyperactive delirium,
7. Patients with chronic kidney disease (CKD, any stage) who received midazolam or morphine infusion during their ICU stay,
8. Patients who received barbiturate coma,
9. Patients who are on theophylline, aminophylline or psychotropic agents at the point of screening for recruitment,
10. Patients with feed intolerant, short bowel syndrome, or
11. Patients with active seizures

Ages: 21 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Duration of mechanical ventilation in days

SECONDARY OUTCOMES:
ICU mortality | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Mortality in the ICU (yes or no)
30-days mortality | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Mortality within 30 days (yes or no)
ICU length of stay | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Length of ICU stay in days
Blood pressure | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Blood pressure in mmHg
Heart rate | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Heart rate in beats per minute
Incidence of arrhythmia | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Incidence of arrhythmia reported (yes or no)
GCS | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Glasgow coma scale
Incidence of re-intubation | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Need for re-intubation following an extubation (yes or no)
Incidence of terminal extubation | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Terminal extubation in the ICU (yes or no)
Need for tracheostomy | From the start of study drug with follow up period of 30 days or until hospital discharge, whichever earlier
  Need for tracheostomy (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon GK Ong, Principal Investigator — A/Professor
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bright M, Raman V, Laupland KB. Use of therapeutic caffeine in acute care postoperative and critical care settings: a scoping review. BMC Anesthesiol. 2021 Mar 31;21(1):100. doi: 10.1186/s12871-021-01320-x. PMID 33789583